CLINICAL TRIAL: NCT06302647
Title: STUDY TO EVALUATE THE WILLINGNESS OF HEALTHY VOLUNTEERS, PATIENTS, DOCTORS AND PHARMACEUTICAL/BIOTECHNOLOGY INDUSTRY TO USE A PLATFORM (WEB OR APP) TO FACILITATE RECRUITMENT AND ENGAGEMENT IN EARLY PHASE CLINICAL TRIALS AND TO IMPROVE THE KNOWLEDGE OF BOTH HEALTHY VOLUNTEERS AND PATIENTS IN CLINCIAL TRIALS
Brief Title: Assessing Interest in Web/App Platforms for Early Phase Clinical Trial Recruitment
Status: Not yet recruiting | Type: Observational
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Responsible Party: Principal Investigator, Paloma Moraga, Project Manager, Instituto de Investigación Hospital Universitario La Paz
Other Study IDs: PI-6022
Record Dates: First submitted 2024-03-04; First posted 2024-03-12 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Assessing Interest in a Platform for Early Phase Clinical Trial Recruitment
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Questionnaire for subjects: Questionnaire will be provided to general subjects anonymously to gain knowledge on their willigness to use a platform to look for early phase clinical trials.
  Interventions: Other: Questionnaires
- Questionnaire for pharma/biotech industry: Questionnaire will be provided to Pharma/biotech industry anonymously to gain knowledge on their willigness to use a platform to promote the recruitment in early phase clinical trials.
  Interventions: Other: Questionnaires
- Questionnaire for doctors: Questionnaire will be provided to Pharma/biotech industry anonymously to gain knowledge on their willigness to use a platform to have information and promote the recruitment in early phase clinical trials.
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Three questionnaires have been developed to be used by subjects, pharmaceutical industry or doctors in regards to the willingness to use a platform for clinical trial recruitment

SUMMARY:
Study objective:

To assess whether the different stakeholders (volunteers, patients, doctors and industry) involved in early phase trials would be interested in using a platform to facilitate recruitment and engagement in this type of trials. In addition, we will also evaluate the degree of awareness existing in society about clinical trials.

Study subjects: General population, patient, physicians, pharmaceutical-biotechnological industry.

Keywords: healthy volunteer, patient, pharma industry, patient associaiton, questionnaire, clinical trial, platform, recruitment, engagement.

ELIGIBILITY:
Inclusion Criteria:

* Participant will be over 18 years old.
* Male, female or do not want to specify.
* Participants will be capable to understand spanish language.
* Subjects able to communicate with the investigator and able to read and write and follow all study instructions.

Exclusion Criteria:

* Individuals not willing to complete the eraly phase clinical trial platform Study survey
* Individuals who do not meet eligibility criteria

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects above 18 years old willing to fulfill the questionnaire
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-03-14 (Estimated); Primary Completion 2024-06-15 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
percentage of each of the three groups that would find the platform useful | 3 months
  It would be deemed useful if they respond affirmatively or, in the case of a numerical scale from 1 to 5 being 1 the worse o low results and 5 the best or highest, if rate it above 4 in 80% of the questions regarding the utility of the platform.